CLINICAL TRIAL: NCT06322706
Title: A Single-Center, Open-Label, Multi-Cycle Study to Evaluate the Pharmacokinetic Profile of Different Doses of ABSK021 Capsules and the Effect of a High-Fat Meal and Omeprazole Enteric-coated Tablets on the Pharmacokinetic Profile of ABSK021 Capsules in Healthy Subjects
Brief Title: A Clinical Trial to Evaluate a High-Fat Meal and Omeprazole Enteric-coated Tablets on ASBK021
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABSK021-105
Record Dates: First submitted 2024-02-29; First posted 2024-03-21 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABSK021 (Experimental)
  Interventions: Drug: ABSK021
- ABSK021and Omeprazole (Experimental)
  Interventions: Drug: ABSK021; Drug: Omeprazole

INTERVENTIONS:
Drug: ABSK021 — ABSK021 oral
Drug: Omeprazole — Omeprazole oral
  Arms: ABSK021and Omeprazole

SUMMARY:
Part A: a single-center, randomized, open-label, three-cycle study to evaluate the pharmacokinetic (PK) profile of different doses of ABSK021 Capsules and the effect of a high-fat meal on the pharmacokinetic profile of ABSK021 Capsules in healthy subjects Part B: a single-center, open-label, fixed-sequence study to evaluate the effect of multiple oral doses of Omeprazole Enteric-coated Tablets on the PK profile of ABSK021 Capsules in healthy subjects

DETAILED DESCRIPTION:
Part A: in this part, 18 healthy subjects are planned to be enrolled and will be randomized to either Study Sequence A (Sequence A) or Study Sequence B (Sequence B) (with 9 subjects in each sequence) to receive single oral dose of ABSK021 separately for a total of 3 doses, separated by 10 days.

Part B: in this part, 18 healthy subjects are planned to be enrolled to receive single oral dose of ABSK021 in a fixed sequence separately for a total of 2 doses. Subjects will receive a single dose of 50 mg ABSK021 Capsules on the morning of Cycle 1 Day 1 (C1D1) under fasting conditions; and 40 mg Omeprazole once daily from Days 1 to 5 of Cycle 2 (C2D1 to C2D5); with the other single oral dose of 50 mg ABSK021 received 2 h after the dose of Omeprazole under fasting conditions on C2D5

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 to 45 years (inclusive) at Screening;
2. Weight ≥ 50.0 kg (male) or ≥ 45.0 kg (female), with a body mass index (BMI) between 19.0 and 28.0 (inclusive), BMI = weight (kg)/height (m)2;
3. Normal or abnormal but not clinically significant results in medical history, physical examination, clinical laboratory tests and other relevant examinations as assessed by the investigator at Screening;
4. Male or female subjects of childbearing potential must agree to use effective methods of contraception during the study and within 6 months after the last dose of investigational product (see section 5.4 for details), and male subjects should not donate sperm during such period; female subjects should not donate ovum during such period and should not be pregnant or lactating. Pregnancy period is defined as the period from the date of conception until termination of pregnancy, and will be determined by laboratory test of human chorionic gonadotropin (hCG) within 7 days prior to initiation of the study;
5. Willing to participate in this study, understand the study procedures and sign the informed consent form prior to screening; willing to comply with the study procedures.

Exclusion Criteria:

1. Past or current medical history of chronic or severe conditions in cardiovascular, respiratory, blood, liver, kidney, gastrointestinal, endocrine or nervous systems;
2. Known or persistent mental disorders that may preclude the subject from participation in the study, as determined by the investigator;
3. Past history of gastric or intestinal surgery, or other operations (except for appendectomy) affecting the drug absorption;
4. Dysphagia and inability to take the investigational product orally;
5. Intolerant to venipuncture, difficult to collect blood samples, and fear of needle sickness and blood;
6. Known allergy to two or more kinds of foods and drugs; or allergic to ABSK021 or its excipients (lactose monohydrate, microcrystalline cellulose, colloidal silicon dioxide, croscarmellose sodium, magnesium stearate, gelatin), allergic to omeprazole; and prone to allergic reactions such as rash and urticaria;
7. History of bacterial, fungal, parasitic, viral (excluding nasopharyngitis), mycobacterial infection, and COVID19 infection within 30 days prior to screening; or abnormal chest X-ray finding, assessed as clinically significant (by the investigator);
8. Symptoms of fatigue and pyrexia within 2 weeks prior to screening;
9. Abnormal laboratory tests: Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 1 × ULN; Creatinine > 1 × ULN; Total Bilirubin (TBIL) > 1.5 × ULN; Creatine Kinase (CK) > 1.5 × ULN; amylase > 1 × ULN; Lactate Dehydrogenase (LDH) > 1.5 × ULN; Serum Potassium < Lower Limit of Normal (LLN); and hemoglobin < LLN;
10. Positive result for either of the following tests: serum Hepatitis B Surface Antigen (HBsAg), Hepatitis B e Antigen (HBeAg), Hepatitis B e Antibody (HBeAb), Hepatitis B Core Antibody (HBcAb), Hepatitis C Virus (HCV) antibody, Human Immunodeficiency Virus (HIV) antibody, and treponema pallidum antibody;
11. Pregnant or lactating women, or those with a positive pregnancy test;
12. Participated in any clinical studies of drugs as a study subject and received the study drug within 3 months prior to screening;
13. Previously participated in any other study related to ABSK021 and received ABSK021;
14. Used strong inhibitors or inducers of CYP3A4 (including grapefruit juice, grapefruit hybrids, punica granatum, carambola, citrus maxima, and Seville oranges [including its juices or other processed products]; see Appendix 12.2Contraindicated Medications and Products for Concomitant Use with ABSK021 or Omeprazole for the detailed list) within 14 days prior to screening and at Screening;
15. Used strong inhibitors or inducers of CYP2C19 (including Fluoxetine, Fluvoxamine, Ticlopidine, Rifampin, etc., see Appendix 12.2 Contraindicated Medications and Products for Concomitant Use with ABSK021 or Omeprazole for the detailed list) within 14 days prior to screening and at Screening;
16. Have special diet requirements and cannot accept to take a unified dietary; specific dietary requirements: (i) the subjects can only eat the food provided by the study site during hospitalization, (ii) the subjects should avoid using strong inhibitors or inducers of CYP3A4 during the study, and (iii) the subjects should avoid using other strong inhibitors or inducers of CYP2C19 during the study (see Appendix 12.2 Contraindicated Medications and Products for Concomitant Use with ABSK021 or Omeprazole for the detailed list);
17. Consumption of more than 14 units of alcohol per week (1 unit of alcohol = about 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 3 months prior to signing the informed consent form, or a positive result for alcohol breath test on the day pre-dose (breath alcohol content > 0.0 mg/100 mL), or unable to abstain from alcohol during the study;
18. Consumption of more than 5 cigarettes per day within 3 months prior to signing the informed consent form, or unable to abstain from tobacco products during the study;
19. Positive for nicotine test;
20. Previous chronic consumption of excessive amount of tea, coffee, or caffeinated beverages (excessive intake is defined as taking more than 6 units of caffeine per day, 1 unit of caffeine equivalent to 177 mL of coffee, 355 mL of tea, 355 mL of cola, or 85 g of chocolate) or unable to abstain from caffeinated beverages during the study;
21. Known history of drug abuse or positive for drug abuse screening test (morphine, methamphetamine, ketamine, methylene dioxyamphetamine, and tetrahydrocannabinol acid);
22. Used over the counter or prescription drugs, including herbal medicine, health products, vitamins, and dietary supplements, within 14 days prior to screening, or plan to use such drugs during the study;
23. Donated or lost > 400 mL of blood within 3 months prior to screening; received blood transfusions or used blood products within 2 months prior to screening;
24. Received vaccine (including COVID19 vaccine) within 2 months prior to screening, or plan to get vaccinated during the study;
25. Significant abnormalities in vital signs, including: ear temperature > 37.7 °C; pulse rate > 100 beats/min or < 50 beats/min; systolic blood pressure ≥ 140 mmHg or < 90 mmHg, diastolic blood pressure ≥ 90 mmHg or < 50 mmHg;
26. Heart rate-corrected QT interval prolongation, QTcF > 450 ms (> 470 ms for females) (Note: QTc interval corrected using the Fridericia formula), or family history of long QT syndrome, or other clinically significant ECG abnormalities at Screening;
27. Plan to donate sperm or ovum within 6 months after administration of the investigational product;
28. Subjects involving in the design or conduct of this study and their immediate family members (e.g., employees of Abbisko Therapeutics Co., Ltd., employees of the CRO, and employees of the study site);
29. Subjects who, in the opinion of the investigator, are not suitable for enrollment or may not be able to complete the study for other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Cmax | predose up to 240 hours post-dose
  PK samples were collected according to the protocol requirements
tmax | predose up to 240 hours post-dose
  PK samples were collected according to the protocol requirements
AUC0-∞ | predose up to 240 hours post-dose
  PK samples were collected according to the protocol requirements
AUClast | predose up to 240 hours post-dose
  PK samples were collected according to the protocol requirements

SECONDARY OUTCOMES:
AE | up to 3 months
  The relationship of each adverse event to the investigational product will be assessed by CTCAE v5.0
SAE | up to 3 months
  The relationship of each serious adverse event to the investigational product will be assessed by CTCAE v5.0
blood pressure | up to 1 months
  blood pressure will be measured by sphygmomanometer
respiratory rate | up to 1 months
  respiratory rate will be measured by respiratory rate machine
ECG QT Interval | predose up to 240 hours post-dose
  12-lead ECGs will be obtained during the study using an ECG machine
t1/2 | predose up to 240 hours post-dose
  PK samples were collected according to the protocol requirements
CL/F | predose up to 240 hours post-dose
  PK samples were collected according to the protocol requirements
Vz/F | predose up to 240 hours post-dose
  PK samples were collected according to the protocol requirements

CONTACTS AND LOCATIONS:
Overall Officials: Kai Huang, Principal Investigator — No. 299, Qingyang Road, Wuxi City, Jiangsu Province
Locations (1):
- Wuxi People's Hospital, Wuxi, JiangShu, China

IPD SHARING:
Plan to Share IPD: No